CLINICAL TRIAL: NCT05365295
Title: Sensitivity of Children With Attention Deficit/Hyperactivity Disorder to Memory Error Production
Brief Title: Study of ADHD Children's Sensitivity to Memory Error Production
Acronym: TDAH-DRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 49RC22-0095
Record Dates: First submitted 2022-04-05; First posted 2022-05-09 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — GREM1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ADHD (Experimental): - ADHD children aged between 8 to 10 years old
  Interventions: Other: DRM (Deese, Roediger et McDermott task)

INTERVENTIONS:
Other: DRM (Deese, Roediger et McDermott task) — Eight lists of nine words are presented to the participants. Each list is heard once. Immediately afterwards, the child is asked to recall the words he or she remembers. Each child's response is then repeated one by one and the participant is asked to rate his or her confidence in the response on a five-point scale (from "not at all sure" to "100% sure"). A 5-minute break is given in the middle of the task, after the first four lists are presented. The test takes about 20 minutes.

SUMMARY:
The purpose of the study is to test whether children with Attention Deficit/Hyperactivity Disorder (ADHD) are more susceptible to false memory production using a DRM paradigm. The number of "critical decoy production" errors will be analyzed and compared to the calibration of the test.

DETAILED DESCRIPTION:
During a neuropsychological assessment, as part of the clinical routine, children with a diagnosis of ADHD, without neurological etiology, aged 8 to 10 years will be offered an additional task. This task, a DRM adapted to the child, consists of learning several lists of words. Each list exposes words belonging to the same lexical field, to a concept not explicitly mentioned in the list, called critical lure. Immediately after the presentation of a list, the child is asked to recall as many words as possible. Recall of the critical lure gives an indication of the production of false memories. The number of critical lures produced by these children will be compared to the calibration of the test, currently being published. The investigator will also verify if the production of critical lures can be correlated with other variables such as performance on intellectual, executive and attentional tasks, proposed during the clinical routine assessment.

The investigator hypothesize that ADHD children will recall more critical lures than the norm, and fewer correct responses than the norm.

The data collected is taken from the child's psychological file. The only personal information used, beyond test performance, is the child's gender and age. The procedure is anonymous.

ELIGIBILITY:
Inclusion Criteria:

* Age between 96 and 131 months
* Child referred by a doctor for a neuropsychological assessment
* Child with ADHD diagnosis
* Sufficient command of the French language
* Non-opposition of the child and his/her parents

Exclusion Criteria:

* Severe psychiatric comorbidity: major depressive episode, bipolar disorder, generalized anxiety disorder, autism spectrum disorder
* Major neurological history: severe head trauma, stroke, severe epilepsy, brain tumor
* Repeating a class during school
* Presence of an intellectual disability
* Use of methylphenidate treatment less than 48 hours before the experiment
* Completion of an intellectual assessment using the Wechsler Intelligence Scale for Children (WISC-V) dated less than one year before the meeting

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
DRM (Deese-Roediger-McDermott task) Performance 1 | 20 minutes during DRM DRM (Deese-Roediger-McDermott) task
  correct answers
DRM (Deese-Roediger-McDermott task) Performance 2 | 20 minutes during DRM DRM (Deese-Roediger-McDermott) task
  critical lures
DRM (Deese-Roediger-McDermott task) Performance 3 | 20 minutes during DRM DRM (Deese-Roediger-McDermott) task
  intruders associated with the lexical field
DRM (Deese-Roediger-McDermott task) Performance 4 | 20 minutes during DRM DRM (Deese-Roediger-McDermott) task
  non-associated intruders
DRM (Deese-Roediger-McDermott task) Performance 5 | 20 minutes during DRM DRM (Deese-Roediger-McDermott) task
  average confidence index for each type of answer

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Martin, Principal Investigator — UH Angers
Locations (2):
- France (2):
  - neuropediatrics department - university hospital center of Angers, Angers
  - Multidisciplinary liberal practice - Acropole Santé, Rezé

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).